CLINICAL TRIAL: NCT02900664
Title: Phase Ib, Open-label, Multi-center Study to Characterize the Safety, Tolerability and Pharmacodynamics (PD) of PDR001 in Combination With CJM112, EGF816, Ilaris® (Canakinumab) or Mekinist® (Trametinib)
Brief Title: A Study of PDR001 in Combination With CJM112, EGF816, Ilaris® (Canakinumab) or Mekinist® (Trametinib)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X2103; 2016-000633-49 (EudraCT Number)
Record Dates: First submitted 2016-05-17; First posted 2016-09-14 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer, Triple Negative Breast Cancer, NSCLC - Adenocarcinoma
Keywords: CRC; TNBC; NSCLC (adenocarcinoma); Immunomodulation; Biomarkers; Bayesian logistic regression model; PDR001; Immunotherapy; Rectal cancer; Metastatic adenocarcinoma; Colorectal cancer; colon cancer; bowel cancer; cancer of the colon and rectum; Colorectal adenocarcinoma; adenocarcinoma; colon; cancer; large intestine; large intestine cancer; colorectum cancer; Triple-negative breast cancer (TNBC); TNBC, basal type; secretory cell; adenoid cystic; medullary; ductal carcinoma; inflammatory; breast carcinoma; breast cancer; breast lump; Pagets disease; HER2 positive metastatic breast cancer; breast cancer positive for human epidermal growth factor receptor 2 (HER2); breast cancer progression; estrogen-receptor (ER) positive(+) breast cancer; Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma; Squamous cell lung carcinoma; Large-cell lung carcinoma; Non small cell lung carcinoma; Non small cell lung cancer; Non-small cell lung cancer; NSCLC; Large cell lung carcinoma; Large cell lung cancer; Pagent's disease
MeSH Terms: conditions — Colorectal Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Rectal Neoplasms; Colonic Neoplasms; Intestinal Neoplasms; Neoplasms; Carcinoma, Ductal; Breast Neoplasms; Lung Neoplasms; Adenocarcinoma of Lung | interventions — spartalizumab; canakinumab; trametinib; nazartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (23):
- PDR + ACZ 100mg Q8W (Experimental): PDR + ACZ 100mg Q8W
  Interventions: Biological: PDR001; Biological: ACZ885
- PDR + ACZ 300mg Q8W (Experimental): PDR + ACZ 300mg Q8W
  Interventions: Biological: PDR001; Biological: ACZ885
- PDR + ACZ RDE TNBC (Experimental): PDR + ACZ Recommended Dose for Expansion (RDE) Triple Negative Breast Cancer (TNBC)
  Interventions: Biological: PDR001; Biological: ACZ885
- PDR + ACZ RDE NSCLC (Experimental): PDR + ACZ Recommended Dose for Expansion (RDE) Non-Small Cell Lung Cancer (NSCLC)
  Interventions: Biological: PDR001; Biological: ACZ885
- PDR + ACZ RDE CRC (Experimental): PDR + ACZ Recommended Dose for Expansion (RDE) Colorectal Cancer (CRC)
  Interventions: Biological: PDR001; Biological: ACZ885
- PDR + CJM 25mg Q4W (Experimental): PDR + CJM 25mg Q4W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + CJM 75mg Q4W (Experimental): PDR + CJM 75mg Q4W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + CJM 225mg Q4W (Experimental): PDR + CJM 225mg Q4W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + CJM 450mg Q4W (Experimental): PDR + CJM 450mg Q4W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + CJM 450mg Q2W (Experimental): PDR + CJM 450mg Q2W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + CJM 900mg Q4W (Experimental): PDR + CJM 900mg Q4W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + CJM 900mg Q2W (Experimental): PDR + CJM 900mg Q2W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + CJM 1200mg Q4W (Experimental): PDR + CJM 1200mg Q4W
  Interventions: Biological: PDR001; Biological: CJM112
- PDR + TMT 0.5mg QD (Experimental): PDR + TMT 0.5mg QD
  Interventions: Biological: PDR001; Drug: TMT212
- PDR + TMT 1mg QD (Experimental): PDR + TMT 1mg QD
  Interventions: Biological: PDR001; Drug: TMT212
- PDR + TMT 1mg QD, 3 Weeks on/1 Week off (Experimental): PDR + TMT 1mg QD, 3 Weeks on/1 Week off
  Interventions: Biological: PDR001; Drug: TMT212
- PDR + TMT 1.5 mg QD, 2 Weeks on/2 Weeks off (Experimental): PDR + TMT 1.5 mg QD, 2 Weeks on/2 Weeks off
  Interventions: Biological: PDR001; Drug: TMT212
- PDR + TMT 1.5 mg QD, 3 Weeks on/1 Week off (Experimental): PDR + TMT 1.5 mg QD, 3 Weeks on/1 Week off
  Interventions: Biological: PDR001; Drug: TMT212
- PDR + EGF816 25mg QD (Experimental): PDR + EGF816 25mg QD
  Interventions: Drug: EGF816
- PDR + EGF816 50mg QD (Experimental): PDR + EGF816 50mg QD
  Interventions: Drug: EGF816
- s.a. ACZ RDE TNBC (Experimental): Single agent (s.a.) ACZ Recommended Dose for Expansion (RDE) Triple Negative Breast Cancer (TNBC)
  Interventions: Biological: ACZ885
- s.a. ACZ RDE NSCLC (Experimental): Single agent (s.a.) ACZ Recommended Dose for Expansion (RDE) Non-Small Cell Lung Cancer (NSCLC)
  Interventions: Biological: ACZ885
- s.a. ACZ RDE CRC (Experimental): Single agent (s.a.) ACZ Recommended Dose for Expansion (RDE) Colorectal Cancer (CRC)
  Interventions: Biological: ACZ885

INTERVENTIONS:
Biological: PDR001 — Powder for solution for infusion
  Other Names: Spartalizumab/PDR001
  Arms: PDR + ACZ 100mg Q8W; PDR + ACZ 300mg Q8W; PDR + ACZ RDE CRC; PDR + ACZ RDE NSCLC; PDR + ACZ RDE TNBC; PDR + CJM 1200mg Q4W; PDR + CJM 225mg Q4W; PDR + CJM 25mg Q4W; PDR + CJM 450mg Q2W; PDR + CJM 450mg Q4W; PDR + CJM 75mg Q4W; PDR + CJM 900mg Q2W; PDR + CJM 900mg Q4W; PDR + TMT 0.5mg QD; PDR + TMT 1.5 mg QD, 2 Weeks on/2 Weeks off; PDR + TMT 1.5 mg QD, 3 Weeks on/1 Week off; PDR + TMT 1mg QD; PDR + TMT 1mg QD, 3 Weeks on/1 Week off
Biological: ACZ885 — Solution for injection
  Other Names: canakinumab
  Arms: PDR + ACZ 100mg Q8W; PDR + ACZ 300mg Q8W; PDR + ACZ RDE CRC; PDR + ACZ RDE NSCLC; PDR + ACZ RDE TNBC; s.a. ACZ RDE CRC; s.a. ACZ RDE NSCLC; s.a. ACZ RDE TNBC
Biological: CJM112 — Solution for infusion
  Arms: PDR + CJM 1200mg Q4W; PDR + CJM 225mg Q4W; PDR + CJM 25mg Q4W; PDR + CJM 450mg Q2W; PDR + CJM 450mg Q4W; PDR + CJM 75mg Q4W; PDR + CJM 900mg Q2W; PDR + CJM 900mg Q4W
Drug: TMT212 — Tablets
  Other Names: trametinib
  Arms: PDR + TMT 0.5mg QD; PDR + TMT 1.5 mg QD, 2 Weeks on/2 Weeks off; PDR + TMT 1.5 mg QD, 3 Weeks on/1 Week off; PDR + TMT 1mg QD; PDR + TMT 1mg QD, 3 Weeks on/1 Week off
Drug: EGF816 — Tablets
  Other Names: Nazartinib
  Arms: PDR + EGF816 25mg QD; PDR + EGF816 50mg QD

SUMMARY:
The purpose of this study was to combine the PDR001 checkpoint inhibitor with each of four agents with immunomodulatory activity to identify the doses and schedule for combination therapy and to preliminarily assess the safety, tolerability, pharmacological and clinical activity of these combinations.

DETAILED DESCRIPTION:
This was a Phase Ib, multi-center, open-label study, to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antitumor activity of PDR001 in combination with canakinumab, CJM112, trametinib and EGF816 and single agent (s.a.) canakinumab in subjects with Triple Negative Breast Cancer (TNBC), Non-Small Cell Lung Cancer (NSCLC) and Colorectal Cancer (CRC). The study comprised a dose escalation part for combination treatments only, followed by a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced/metastatic cancer, with measurable disease as determined by RECIST version 1.1, who have progressed despite standard therapy or are intolerant to standard therapy, and for whom no effective therapy is available.

Patients must fit into one of the following groups:

* Colorectal cancer (CRC) (not mismatch repair deficient by local assay including PCR and/or immunohistochemistry)
* Non-small cell lung cancer (NSCLC) (adenocarcinoma)
* Triple Negative Breast Cancer (TNBC) (D
* ECOG Performance Status ≤ 2
* Patient must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at baseline, and again during therapy on this study.
* Prior therapy with PD-1/PDL-1 inhibitors is allowed provided any toxicity attributed to prior PD-1- or PD-L1-directed therapy did not lead to discontinuation of therapy.
* Written informed consent must be obtained prior to any screening procedures other than procedures performed as part of standard of care.

Exclusion Criteria:

* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy, or increasing doses of corticosteroids within the prior 2 weeks.
* History of severe hypersensitivity reactions to other monoclonal antibodies.
* Out of range laboratory values for measures of hepatic and renal function, electrolytes and blood counts
* Impaired cardiac function or clinically significant cardiac disease.
* Patients with active, known or suspected autoimmune disease.
* Human Immunodeficiency Virus infection at screening.
* Escalation part: Active Hepatitis B (HBV) or Hepatitis C (HCV) virus infection at screening.

Expansion part: Patients with active HBV or HCV are excluded, excepting those patients undergoing treatment for HBV or HCV.

* Malignant disease, other than that being treated in this study.
* Recent systemic anti-cancer therapy
* Active infection requiring systemic antibiotic therapy.
* Patients requiring chronic treatment with systemic steroid therapy, other than replacement dose steroids in the setting of adrenal insufficiency or treatment with low, stable dose of steroid (<10mg/ day prednisone or equivalent) for stable CNS metastatic disease.
* Patients receiving systemic treatment with any immunosuppressive medication, excepting the above
* Use of any live vaccines against infectious diseases (e.g. influenza, varicella, pneumococcus) within 4 weeks of initiation of study treatment.
* Participation in an interventional, investigational study within 2 weeks of the first dose of study treatment.
* Presence of ≥ CTCAE grade 2 toxicity (except alopecia and ototoxicity, which are excluded if ≥ CTCAE grade 3) due to prior cancer therapy.
* Recent use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GMCSF, M-CSF)

Additional exclusion criteria for Combination arm PDR001+canakinumab and single-agent canakinumab

* Patients with tuberculosis (TB). Note: Patient with latent TB may be eligible based on the investigator's benefit-risk assessment.
* Patients who have been infected with HBV or HCV including those with inactive disease.

Additional exclusion criteria for Combination arm PDR001+CJM112

* Patients with TB. Note: Patient with latent TB may be eligible based on the investigator's benefit-risk assessment.
* Patients with history of and/or active inflammatory bowel disease.
* Active skin or soft tissue infection including cellulitis, erysipelas, impetigo, furuncle,carbuncle, abscess, or fasciitis.
* Active candida infection, including mucocutaneous infection or history of invasive candidiasis.

Additional exclusion criteria for Combination arm PDR001+trametinib

* Patients with history of retinal vein oclusion.
* Patients with history of interstitial lung disease or pneumonitis.
* Patients with cardiomyopathy and/or LVEF < LLN.
* Impairment of gastrointestinal function or GI disease that may significantly alter the absorption of oral combination partners.
* Hemoglobin (Hgb) < 9 g/dL without growth factor or transfusion support
* Women of child-bearing potential using hormonal contraception, unless an additional contraception method is also used according to the Mekinist® label.

Additional exclusion criteria for Combination arm PDR001+EGF816

* NSCLC patients with EGFR mutant tumors.
* Strong inhibitors and strong inducers of CYP3A4 should not be used concomitantly.
* Patients with history of interstitial lung disease.
* Patients who have been infected with HBV or HCV including those with inactive disease.
* Impairment of gastrointestinal function or GI disease that may significantly alter the absorption of oral combination partners
* Patients cannot have received radiotherapy to lung fields within 6 months of study treatment start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) as a measure of safety | Throughout the study at every visit, an average of 1 year
Changes between baseline and post-baseline laboratory parameters and vital signs. | Baseline and throughout the study at every visit, an average of 1 year
Incidence of dose limiting toxicities (DLTs) of treatment (Escalation only) | During the first two cycles; Cycle = 28 days
Frequency of dose interruptions | Throughout the study at every visit, an average of 1 year
Dose intensities | Throughout the study at every visit, an average of 1 year
Severity of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) as a measure of safety | Throughout the study at every visit, an average of 1 year
Frequency of dose reductions | Throughout the study at every visit, an average of 1 year

SECONDARY OUTCOMES:
Key secondary: Histopathology of tumor infiltrating lymphocytes (TILs) | Baseline and approximately after 2 cycles of treatment and at disease progression; Cycle = 28 days
Changes from baseline in electrocardiogram (ECG) parameters | Baseline and end of treatment, an average of 1 year
Best overall response (BOR) | T1: Every 2 cycles until the start of T2. T2: Every 2 cycles until cycle 3 and then every 3 cycles until PD; cycle = 28 days
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Progression free survival (PFS) per irRC and RECIST v1.1 | T1: Every 2 cycles until the start of T2. T2: Every 2 cycles until cycle 3 and then every 3 cycles until PD; cycle = 28 days
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Treatment Free Survival (TFS) | T1: Every 2 cycles until the start of T2. T2: Every 2 cycles until cycle 3 and then every 3 cycles until PD; cycle = 28 days
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Presence and/or concentration of anti-PDR001 antibodies. | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Serum concentration of PDR001, canakinumab, CJM112 | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Plasma concentrations of trametinib and EGF816 | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Key secondary: Histopathology of myeloid cell infiltrate by IHC (such as CD8, FoxP3 and myeloid markers as appropriate). | Baseline and approximately after 3 cycles of treatment and at disease progression; cycle = 28 days
PK parameters (Eg. TMax) of EGF816 | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
PK parameters (Eg. TMax) of trametinib | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
PK parameter (Eg. TMax) of PDR001 | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
PK parameters (Eg. TMax) of canakinumab | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
PK parameters (Eg. TMax) of CJM112 | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Presence and/or concentration of anti-canakinumab antibodies. | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2
Presence and/or concentration of anti-CJM112 antibodies. | Cycle 1 through cycle 6 in treatment period 1 and 2 (an average of 1 year)
  T1: treatment period 1 (6 cycles of treatment) T2: treatment period 2

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (4):
  - Sidney Kimmel Comprehensive Cancer Center SC-3, Baltimore, Maryland
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Wilrijk
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (4):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CPDR001X2103 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17917